CLINICAL TRIAL: NCT03584750
Title: Floating for Chronic Pain (Float4Pain)
Brief Title: Floating for Chronic Pain
Acronym: Float4Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hannover Medical School (Other)
Responsible Party: Principal Investigator, Beißner, Florian Prof. Dr., Principal Investigator, Hannover Medical School
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 7684
Record Dates: First submitted 2018-06-11; First posted 2018-07-12 (Actual); Last update posted 2020-11-24 (Actual); Status verified 2020-11

CONDITIONS: Chronic Pain Syndrome
Keywords: Somatic and psychological factors
MeSH Terms: interventions — Divorce

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention group (Active Comparator): Floating
  Interventions: Other: Floating
- Control group (Placebo Comparator): Placebo floating
  Interventions: Other: Placebo floating
- No-treatment group (No Intervention): Waiting list

INTERVENTIONS:
Other: Floating — Floating in specialized tank with full floatation and sensory deprivation.
  Other Names: Floatation REST
  Arms: Intervention group
Other: Placebo floating — Floating in specialized tank with reduced floatation and sensory deprivation.
  Arms: Control group

SUMMARY:
In recent years there has been a novel approach for the treatment of chronic pain: Floatation REST (restricted environmental stimulation therapy). Floating is a therapeutic approach, in which patients float in a specialized pool or tank on water that contains high concentrations of Epsom salt (Magnesium sulfate). Water is kept at skin temperature (35-36°C) and the pool or tank is shielded to provide almost complete darkness and silence. This therapeutic approach has proven to be effective in alleviating chronic pain.

Due to the difficulties associated with designing a credible placebo control there have been no randomized controlled trials (RCTs) with patients blinding so far. Such blinding, however, is crucial, to assess the true therapeutic effect of the intervention.

The investigators will conduct the first patient blinded RCT of Floatation REST for chronic pain with a credible placebo control for floating and a no-treatment group.

ELIGIBILITY:
Inclusion Criteria:

* Current diagnosis of chronic pain disorder with somatic and psychological factors (German ICD F45.41)
* Able and willing to give written informed consent

Exclusion Criteria:

* Pregnant or nursing women (self report)
* Previous experience with floating
* Acute illnesses that may exacerbate or shadow the chronic pain condition (acute inflammation, major depression, active neoplasm, etc.)
* History of alcohol and drug abuse
* Any clinically relevant abnormal findings in the clinical history, which, in the opinion of the investigator, may either put the subject at risk because of participation in the study or may influence the results of the study or the subject's ability to participate in the study.
* Any clinical condition that may prevent the subject from floating, such as: open injuries, contagious diseases (influenza, GI infections, athlete's foot), GERD, epilepsy, claustrophobia, schizophrenia, incontinence or acute skin disorders.
* Suspected inability to understand the protocol requirements, instructions and study-related restrictions, the nature, scope, and possible consequences of the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2018-06-26 (Actual); Primary Completion 2020-01-02 (Actual); Study Completion 2020-06-18 (Actual)

PRIMARY OUTCOMES:
Change in Pain intensity (maximum and average) as compared to baseline | 1, 12 and 24 weeks after intervention
  Numeric rating scales from 0 ("no pain") to 100 ("maximum imaginable pain"), assessing retrospectively the week before.

SECONDARY OUTCOMES:
Change in Pain scores (maximum and average, dichotomous) as compared to baseline | 1, 12 and 24 weeks after intervention
  Numeric rating scale from 0 ("no pain") to 100 ("maximum imaginable pain"), assessing retrospectively the week before. A change of 30% or more pain reduction will be considered a success.
Change in pain-related disability as compared to baseline | 1, 12 and 24 weeks after intervention
  Pain related disability will be assessed via the Pain Disability Index (PDI). The total score ranges from 0 (no pain-related disability) to 70 (maximal disability).
Change in trait anxiety as compared to baseline | 1, 12 and 24 weeks after intervention
  Trait anxiety will be assessed via the "State-Trait Anxiety Inventory (STAI) Form X2". The total score ranges from 20 to 80, with higher scores indicating greater anxiety.
Change in depression as compared to baseline | 1, 12 and 24 weeks after intervention
  Depression will be assessed via the Becks Depression Inventory (BDI). The total score ranges from 0 (no depression) to 63 (severe depression).
Change in physical and mental health as compared to baseline | 1, 12 and 24 weeks after intervention
  This will be assessed via the "12-Item Short Form Survey (SF-12v2)". This questionnaire yields two scores that will be reported separately: Physical Component Summary (PCS) and Mental Component Summary (MCS), both normalised to 50 with a standard deviation of 10. Where values larger than 50 represent better than average health.
Change in quality of sleep assessed by a numeric rating scale as compared to baseline | 1, 12 and 24 weeks after intervention
  Participants will be asked how much their pain impairs their sleep on a scale from 0 ("not at all") to 100 ("very much").
Change in use of pain medication as compared to baseline | 1, 12 and 24 weeks after intervention
  Self reported list
Change in pain area as compared to baseline | 1 week after intervention
  Pain area derived from electronic pain drawings (SymptomMapper). Pain area ranges from 0 to 100% of body area.
Change in pain widespreadness as compared to baseline | 1 week after intervention
  Widespread pain index (WPI) derived from electronic pain drawings (SymptomMapper). The WPI ranges from 1 (pain localised in one region) to 19 (pain affects all possible regions).
Change in pain intensity | Immediately before - immediately after every float session
  Same as Outcome 1, but for acute pain
Change in pain area and widespreadness | Immediately before - immediately after every float session
  Same as Outcome 9, but for acute pain
Change in state anxiety | Immediately before - immediately after every float session
  State anxiety will be assessed via the "State-Trait Anxiety Inventory (STAI) Form X1". Scores range from 20 to 80, with higher scores indicating greater anxiety.
Change in heart rate | Immediately before - immediately after every float session
  Heart rate [bpm] will be derived from a 5-minute ECG recording. Normative values range between 60 and 90 bpm.
Change in high frequency (HF) power of heart rate | Immediately before - immediately after every float session
  HF power (0.15-0.4 Hz) will be derived from a 5-minute ECG recording. Normative values range between 770-1078 ms^2.
Change in low frequency (LF) power of heart rate | Immediately before - immediately after every float session
  LF power (0.04-0.15 Hz) will be derived from a 5-minute ECG recording. Normative values range between 754-1078 ms^2.
Change in the LF/HF ratio of heart rate | Immediately before - immediately after every float session
  See outcomes 15 and 16 for LF and HF frequency bands. Normative values range between 1.5-2.
Change in the standard deviation of NN intervals (SDNN) | Immediately before - immediately after every float session
  SDNN [ms] will be derived from a 5-minute ECG recording. Normative values range between 30-100 ms.
Change in the root mean square of successive differences (RMSSD) | Immediately before - immediately after every float session
  RMSSD [ms] will be derived from a 5-minute ECG recording. Normative values range between 15-45 ms.
Change in the coefficient of variation (CV) | Immediately before - immediately after every float session
  CV [%] will be derived from a 5-minute ECG recording. Normative values range between 3-12%.
Change in the proportion of NN50 divided by total number of NNs (pNN50) | Immediately before - immediately after every float session
  pNN50 [%] will be derived from a 5-minute ECG recording. Normative values range between 15-34%.
Unusual bodily sensations during floating | During floating
  Electronic drawing
Change in relaxation | Immediately before - immediately after every float session
  Relaxation will be assessed via numeric rating scale from 0 ("not relaxed at all") to 100 ("completely relaxed").

CONTACTS AND LOCATIONS:
Overall Officials: Florian Beissner, Dr. phil. nat., Principal Investigator — Hannover Medical School
Locations (1):
- Hannover Medical School, Hanover, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Loose LF, Manuel J, Karst M, Schmidt LK, Beissner F. Flotation Restricted Environmental Stimulation Therapy for Chronic Pain: A Randomized Clinical Trial. JAMA Netw Open. 2021 May 3;4(5):e219627. doi: 10.1001/jamanetworkopen.2021.9627. PMID 33988708